CLINICAL TRIAL: NCT05248958
Title: Turkish Adaptation, Validity and Reliability of Cravings for Rest and Volitional Energy Expenditure (CRAVE)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, research assistant, Istanbul Medeniyet University
Other Study IDs: CRAVE
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-06

CONDITIONS: Exercise; Motivation; Sedantary Activity
Keywords: exercise; motivation; physical activity; sedantary activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Turkish Validity and Reliability of The CRAVE Scale — The aim of this study is to adapt the Cravings for Rest and Volitional Energy Expenditure (CRAVE) scale to Turkish society and to make its validity and reliability in Turkish.

SUMMARY:
The aim of this study is to adapt the Cravings for Rest and Volitional Energy Expenditure (CRAVE) scale to Turkish society and to make its validity and reliability in Turkish. The CRAVE scale developed by Stults-Kolehmainen et al assesses the intrinsic motivation required for sedentary behavior and participation in physical activity. It has 13 questions. CRAVE scale questions and questions in the data collection form will be prepared through the google surveys and will be sent to the participants via Whatsapp, Facebook, Instagram and e-mail. Participants will fill out the survey forms online. 130 participants will be included in the study. In order to evaluate the validity of the CRAVE, the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2), which can measure exercise behaviors and intrinsic motivation and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

DETAILED DESCRIPTION:
The reliability and validity of the scale will begin with language equivalence and cultural adaptation. The scale will be translated from English to Turkish by two people who are fluent in Turkish and English. A single Turkish translation will be obtained from these two Turkish translations with a common opinion. The scale, which has been translated into Turkish, will be translated into English by two other people who are fluent in Turkish and English. The scale translated into English will be compared with the original. If the developer of the scale, miguel blacutt and Stults-Kolehmainen approves the translation of the scale, participants will be recruited for the study. In the pre-trial phase, a pre-assessment will be conducted with 15 participants to test the intelligibility of the scale. Based on the results of the pre-test phase, the final version of CRAVE will be able to be modified. RAVE scale questions and questions in the data collection form will be prepared through the google surveys and will be sent to the participants via Whatsapp, Facebook, Instagram and e-mail. Participants will fill out the survey forms online. 130 participants will be included in the study. In order to evaluate the validity of the CRAVE, the Behavioral Regulation in Exercise Questionnaire-2 (BREQ-2), which can measure exercise behaviors and intrinsic motivation and has been validated in Turkish, will be used. Scales will be repeated after 15 days to assess test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-30 years
* Adult individuals who have access to the Internet and agreed to participate in the study. -
* Native language being Turkish

Exclusion Criteria:

* Inability to use a computer, tablet or mobile phone
* Native language not being Turkish

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: - Persons who meet the inclusion criteria and who volunteered to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
exercise motivation | baseline
  Exercise motivation will be assessed with CRAVE scale. It consists of 13 items in total. Each item is scored on a scale of 0-10, ranging from "never" to "more than ever". The scale includes two sub-categories: "rest motivation" and "intrinsic motivation to move". There are 5 questions in the resting category and 5 questions in the moving category, and 3 questions are not scored. The score of each category is calculated by dividing the total score of the questions in that category by the number of questions.
exercise behaviour | baseline
  Exercise behaviour will be assessed with BREQ-2 Scale. It comprises 19 items with ratings on a 5-point Likert scale ranging from 0 (not true for me) to 4 (very true for me). It measures amotivated (e.g., "I think exercising is a waste of time"), external (e.g., "I exercise because other people say I should"), introjected (e.g., "I feel guilty when I don't exercise"), identified (e.g., "it's important to me to exercise regularly"), and intrinsic (e.g., "I find exercise a pleasurable activity") regulations of exercise behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided